CLINICAL TRIAL: NCT06767982
Title: A Randomized Prospective Trial Comparing Bacillus Calmette-Guerin (BCG) RIVM and Russian Strains in Non-Muscle Invasive Bladder Cancer: Efficacy and Side Effects
Brief Title: Comparison of BCG RIVM and Russian Strains for Treating Non-Muscle-Invasive Bladder Cancer (NMIBC)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Khaled Obaid, Principal Investigator , Urologist, Ankara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: İ10-640-21
Record Dates: First submitted 2024-12-26; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Non Muscle Invasive Bladder Cancer
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms | interventions — BCG Vaccine

STUDY DESIGN:
Intervention Model Description: This randomized, prospective trial included 125 patients with intermediate-, high-, and very high-risk non muscle invasive bladder cancer. Patients were randomized into two groups to receive either the BCG RIVM or BCG Russian substrain following transurethral resection of bladder tumor (TURBT).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 which received BCG RIVM (Active Comparator): following transurethral resection of bladder tumor (TURBT), patients in Group 1 received BCG RIVM.
  Interventions: Drug: Bacillus Calmette-Guerin (BCG)
- Group 2 which received BCG RUSSIAN (Active Comparator): following transurethral resection of bladder tumor (TURBT), patients in Group 2 received BCG RUSSIAN.
  Interventions: Drug: Bacillus Calmette-Guerin (BCG)

INTERVENTIONS:
Drug: Bacillus Calmette-Guerin (BCG) — In this study we compared the efficacy and side effects of two different strains of BCG (RIVM and RUSSIAN strains) in non muscle invasive bladder cancer patients

SUMMARY:
The goal of this clinical trial is to compare the efficacy and safety of two Bacillus Calmette-Guérin (BCG) substrains (RIVM and Russian) in the treatment of intermediate- and high-risk non-muscle-invasive bladder cancer (NMIBC) in adult patients.

The main questions it aims to answer are:

* Is there a significant difference in recurrence-free survival (RFS) between the BCG RIVM and BCG Russian substrains?
* Is there a significant difference in progression-free survival (PFS) between the two substrains?
* Are there notable differences in the incidence of treatment-related adverse events between the strains? Researchers will compare patients treated with BCG RIVM to patients treated with BCG Russian to determine whether one substrain offers superior clinical outcomes in terms of recurrence, progression, and adverse events.

Participants will:

Undergo transurethral resection of bladder tumor (TURBT) prior to initiating therapy.

Be randomly assigned to receive either BCG RIVM or BCG Russian intravesical therapy.

Receive an induction course of six weekly instillations of the assigned BCG substrain.

Receive maintenance therapy at regular intervals (3, 6, 12, 18, 24, 30, and 36 months) based on risk classification.

Undergo regular follow-up with cystoscopy and urine cytology to assess recurrence, progression, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years,
* histopathologically confirmed NMIBC (stages Ta, T1, or CIS),
* classification as intermediate, high, or very high risk (who either refused or were not suitable candidates for radical cystectomy),
* no prior BCG therapy,
* no evidence of upper urinary tract carcinoma or distant metastases and
* a minimum follow-up period of 12 months.

Exclusion Criteria:

* patients who did not receive adequate BCG therapy (defined as receiving fewer than 5 of the 6 induction doses or fewer than 2 of the 3 maintenance doses),
* patients with a follow-up period of less than 12 months and
* patients who received multiple BCG strains during the follow-up period.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
recurrence free survival | Through study completion, up to 4 years
progression free survival | Through study completion, up to 4 years

SECONDARY OUTCOMES:
side effects of the treatment | At each BCG instillation and follow-up visit, up to 4 years

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University Faculty of Medicine Ibni Sina Hospital, Ankara, Altindag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Unda-Urzaiz M, Cozar-Olmos JM, Minana-Lopez B, Camarero-Jimenez J, Brugarolas-Rossello X, Zubiaur-Libano C, Ribal-Caparros MJ, Suarez-Charneco AJ, Rodriguez-Tesedo V, Chantada-Abal V, Ruiz-de-Leon C, Carrillo-George C, Carballido-Rodriguez J, Villacampa-Auba F; en representacion del Grupo Espanol del Registro de Cepas de BCG. Safety and efficacy of various strains of bacille Calmette-Guerin in the treatment of bladder tumours in standard clinical practice. Actas Urol Esp (Engl Ed). 2018 May;42(4):238-248. doi: 10.1016/j.acuro.2017.10.003. Epub 2017 Dec 30. English, Spanish. PMID 29295749
- [Background] Niwa N, Kikuchi E, Matsumoto K, Kosaka T, Mizuno R, Oya M. Does switching the bacillus Calmette-Guerin strain affect clinical outcome in patients with recurrent non-muscle-invasive bladder cancer after initial bacillus Calmette-Guerin therapy? Urol Oncol. 2018 Jun;36(6):306.e1-306.e8. doi: 10.1016/j.urolonc.2018.02.005. Epub 2018 Mar 9. PMID 29530465
- [Background] Krajewski W, Matuszewski M, Poletajew S, Grzegrzolka J, Zdrojowy R, Kolodziej A. Are There Differences in Toxicity and Efficacy between Various Bacillus Calmette-Guerin Strains in Bladder Cancer Patients? Analysis of 844 Patients. Urol Int. 2018;101(3):277-284. doi: 10.1159/000492722. Epub 2018 Sep 18. PMID 30227437
- [Background] Del Giudice F, Busetto GM, Gross MS, Maggi M, Sciarra A, Salciccia S, Ferro M, Sperduti I, Flammia S, Canale V, Chung BI, Conti SL, Eisenberg ML, Skinner EC, De Berardinis E. Efficacy of three BCG strains (Connaught, TICE and RIVM) with or without secondary resection (re-TUR) for intermediate/high-risk non-muscle-invasive bladder cancers: results from a retrospective single-institution cohort analysis. J Cancer Res Clin Oncol. 2021 Oct;147(10):3073-3080. doi: 10.1007/s00432-021-03571-0. Epub 2021 Mar 6. PMID 33675400
- [Background] Huang Z, Liu H, Wang Y, Zhang C, Xu T. Determining optimal maintenance schedules for adjuvant intravesical bacillus Calmette-Guerin immunotherapy in non-muscle-invasive bladder cancer: a systematic review and network meta-analysis. Curr Med Res Opin. 2017 Aug;33(8):1379-1387. doi: 10.1080/03007995.2017.1326889. Epub 2017 Jun 6. PMID 28471272

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-01-01): https://cdn.clinicaltrials.gov/large-docs/82/NCT06767982/Prot_SAP_000.pdf